CLINICAL TRIAL: NCT06278103
Title: Correlation Between Expression of Hormonal Receptors, Clinical Data, and Methylation Profile in Meningiomas
Brief Title: Correlation Between Expression of Hormonal Receptors, Clinical Data, and Methylation Profile in Meningiomas (MethylRH-M)
Acronym: MethylRH-M
Status: Enrolling by invitation | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Guillaume GAUCHOTTE, Professor, Central Hospital, Nancy, France
Other Study IDs: 2023PI113
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Meningioma
Keywords: Meningioma; Hormonal receptors
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Years
Biospecimen Retention: Samples With DNA — FFPE blocks. Frozen tumoral tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research aims to explore the relationship between hormonal receptor expression and the clinical and histopathological characteristics of meningiomas. The underlying hypothesis is that hormonal receptor expression, as well as the methylation profile of their gene promoters, are associated with specific aspects of meningiomas and patients' clinical outcomes. The main objective is to study the correlation between the immunohistochemical expression of hormonal receptors and clinicopathological data. The secondary objectif is to study the correlation between the methylation profile of hormonal receptor gene promoters and their immunohistochemical expression.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery for a meningioma at the University Hospital of Nancy between 2000 and 2022.

Exclusion Criteria:

* Patients who did not express their consent to participate in the study.
* Patients with grade 2 or 3 meningiomas whose samples are no longer available or in insufficient quantity to perform an immunohistochemical study.
* Patients with grade 1 meningiomas not selected by randomization.
* Patients withdrawing their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgery for a meningioma at the University Hospital of Nancy between 2000 and 2022.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
immunohistochemical expression of different hormonal receptors | up to 24 years after surgery
  Evaluated on FFPE sections

SECONDARY OUTCOMES:
methylation profile of the promoters of hormonal receptor genes | up to 24 years after surgery
  Methylation profile established from frozen tissue.

IPD SHARING:
Plan to Share IPD: Undecided